CLINICAL TRIAL: NCT02895698
Title: Effects of Myofascial Trigger Point Dry Cupping on Plantar Heel Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2014-04-322
Record Dates: First submitted 2016-09-06; First posted 2016-09-12 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Plantar Fasciitis; Heel Spur Syndrome; Chronic Plantar Fasciitis
Keywords: Cupping; Dry cupping; Myofascial trigger points
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Active Comparator): Dry cupping + active dorsiflexion exercise + stretching exercise
  Interventions: Device: Dry cupping
- Control group (Other): stretching exercise + active dorsiflexion without cupping
  Interventions: Other: Stretching exercises

INTERVENTIONS:
Device: Dry cupping — Dry cupping. First, the therapist identified the trigger point on calf muscle.After identification of the trigger point, the participant was in prone with the ankle outside the edge of the bed. Ultrasound gel was then placed over the trigger point as a lubricant to increase the suctioning of the plastic vacuum cup, after which the cup was placed. Air was withdrawn from the cup to create a suction force. The cup was maintained for 10 minutes, and the participant was asked to do active ankle dorsiflexion exercise after 5 minutes of placing the cup. The therapist held the cup in place while the participant performed exercise.
  Arms: Treatment group
Other: Stretching exercises — * The participant was in prone with the ankle outside the edge of the bed. The participant was asked to do active ankle dorsiflexion exercise after 5 minutes of lying on bed.
  * Standing self-stretching of the calf muscles.
  * Plantar fascia-specific self-stretching.The participant was instructed to start gently at first and then to work more aggressively as long as the pain is tolerable.
  * All stretches were done six times and the duration of each stretch is 30 seconds.
  Arms: Control group

SUMMARY:
The main aim of this study is to investigate the effects of dry cupping on calf muscle trigger points in patients with plantar heel pain. A secondary aim is to examine the correlation between several outcome measures in those patients.

DETAILED DESCRIPTION:
Plantar heel pain is a condition often seen by healthcare providers. It is presented as pain and tenderness under the heel with weight bearing activities. Approximately 15% of athletic and non-athletic adults who have foot complaints seek professional care for plantar heel pain. There are different names and definitions for this condition in the literature such as plantar heel pain, plantar fasciitis, plantar fasciosis, plantar fasciopathy, heel spur syndrome, and jogger's heel. The reason for inconsistency in defining the condition is due to disagreement on the underlying pathology. A number of conditions may result in plantar heel pain, namely plantar fasciitis (most common), calcaneus fracture, heel fat pad atrophy, and peripheral nerve dysfunction. Recently, several studies have shown that myofascial trigger points (MTrPs) or tender points in the calf muscles may be associated with plantar heel pain. Many studies have determined risk factors in the development of plantar heel pain, classifying them as either intrinsic or extrinsic. Intrinsic risk factors comprise the anatomical (ROM of the ankle and subtalar joints position) or demographic characteristics of the individual (age, gender, weight and height). Extrinsic risk factors are related mainly to the subject's activity environment, such as running on a hard surface, time spent weight bearing, and previous injury. All these factors lead to an increase in the mechanical load on the foot, specifically the plantar fascia. Treatment of plantar heel pain usually targets the plantar fascia or other structures in the plantar heel area using several interventions such as cortisone injection, therapeutic ultrasound, laser, ice, heel pads, and night splints. Evidence varies regarding the effectiveness of these interventions.

The main aim of this study is to investigate the immediate and carry-over effects of dry cupping on calf muscle trigger points on pain and function in patients with plantar heel pain.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral plantar heel pain.
* Trigger point(s) in the gastrocnemius/soleus muscle(s).
* Central or centro-medial tenderness in the plantar aspect of the heel.

Exclusion Criteria:

* Red flags: tumor, fracture, rheumatoid arthritis, osteoporosis, or any severe vascular condition in the lower limbs.
* Neurological symptoms: sciatica, tarsal tunnel syndrome.
* Previous surgery in the affected leg below the hip.
* Fibromyalgia.
* Previous manual therapy treatment for the same condition within the past 6 months.
* History of more than three corticosteroid injections within the past year.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | Change from Baseline in VAS at 5 minutes post intervention
  * A self-reporting scale.
  * The scale is presented as a 10-cm horizontal line on which the participant pain intensity is represented by a point between the two ends: one end is labelled no pain, and the other end is labelled worst pain imaginable.
Visual analogue scale (VAS) | Change from Baseline in VAS at 2 days post intervention
  * A self-reporting scale.
  * The scale is presented as a 10-cm horizontal line on which the participant pain intensity is represented by a point between the two ends: one end is labelled no pain, and the other end is labelled worst pain imaginable.
Morning first steps visual analogue scale | Change from Baseline in morning visual Analog Scale at 2 days post intervention
  * A self-reporting scale.
  * The scale is presented as a 10-cm horizontal line on which the participant pain intensity is represented by a point between the two ends: one end is labelled no pain, and the other end is labelled worst pain imaginable.
Pressure pain threshold (PPT) | Change from Baseline in PPT at 5 minutes post intervention
  * The PPT was measured with an electronic algometer.
  * Pressure was applied at a rate of 40 kilopascal (kPa/s), and participants pressed a switch when the sensation changed from pressure only to pressure and pain.
Pressure pain threshold (PPT) | Change from Baseline in PPT at 2 days post intervention
  * The PPT was measured with an electronic algometer.
  * Pressure was applied at a rate of 40 kPa/s, and participants pressed a switch when the sensation changed from pressure only to pressure and pain.
The patient-specific functional scale (PSFS) | Change from Baseline in PSFS at 2 days post intervention
  * A clinical outcome measure that allows participant to state their own functional status.
  * The examiner asked the participant about three important activities that they were unable to do or had difficulty doing. The participants rated their level of function on a scale starting from 0, which is the lowest functional level, and 10, which is the highest level of function.
Ankle dorsiflexion range of motion (ROM) | Change from Baseline in ankle dorsiflexion ROM at 5 minutes post intervention
  * An inclinometer was used to measure the ROM of ankle dorsiflexion.
  * The participant stands in a calf-stretch position, with knee extended or knee flexed (modified lunge position) then to move forward until the heel starts to rise or to maximum stretch. Then the examiner measured the range of motion.
Ankle dorsiflexion range of motion (ROM) | Change from Baseline in ankle dorsiflexion ROM at 2 days post intervention
  * An inclinometer was used to measure the ROM of ankle dorsiflexion.
  * The participant stands in a calf-stretch position, with knee extended or knee flexed (modified lunge position) then to move forward until the heel starts to rise or to maximum stretch. Then the examiner measured the range of motion.
Ankle plantar flexion strength | Change from Baseline in ankle plantar flexion strength at 5 minutes post intervention
  Ankle plantar flexion strength was assessed by asking the participant to perform as many single-leg heel rises as possible in standing at a rate of one every 2 seconds, and the examiner counted the repetitions.
Ankle plantar flexion strength | Change from Baseline in ankle plantar flexion strength at 2 days post intervention
  Ankle plantar flexion strength was assessed by asking the participant to perform as many single-leg heel rises as possible in standing at a rate of one every 2 seconds, and the examiner counted the repetitions.

CONTACTS AND LOCATIONS:
Overall Officials: Ali M Al Shami, Ph.D, Study Director — Imam Abdulrahman Bin Faisal University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crawford F, Thomson C. Interventions for treating plantar heel pain. Cochrane Database Syst Rev. 2003;(3):CD000416. doi: 10.1002/14651858.CD000416. PMID 12917892
- [Background] Radford JA, Landorf KB, Buchbinder R, Cook C. Effectiveness of calf muscle stretching for the short-term treatment of plantar heel pain: a randomised trial. BMC Musculoskelet Disord. 2007 Apr 19;8:36. doi: 10.1186/1471-2474-8-36. PMID 17442119
- [Background] Ieong E, Afolayan J, Carne A, Solan M. Ultrasound scanning for recalcitrant plantar fasciopathy. Basis of a new classification. Skeletal Radiol. 2013 Mar;42(3):393-8. doi: 10.1007/s00256-012-1470-x. Epub 2012 Jul 22. PMID 22820618
- [Background] Irving DB, Cook JL, Menz HB. Factors associated with chronic plantar heel pain: a systematic review. J Sci Med Sport. 2006 May;9(1-2):11-22; discussion 23-4. doi: 10.1016/j.jsams.2006.02.004. Epub 2006 Apr 3. PMID 16584917
- [Background] Alshami AM, Souvlis T, Coppieters MW. A review of plantar heel pain of neural origin: differential diagnosis and management. Man Ther. 2008 May;13(2):103-11. doi: 10.1016/j.math.2007.01.014. Epub 2007 Mar 30. PMID 17400020
- [Background] Messier SP, Pittala KA. Etiologic factors associated with selected running injuries. Med Sci Sports Exerc. 1988 Oct;20(5):501-5. PMID 3193867
- [Background] Renan-Ordine R, Alburquerque-Sendin F, de Souza DP, Cleland JA, Fernandez-de-Las-Penas C. Effectiveness of myofascial trigger point manual therapy combined with a self-stretching protocol for the management of plantar heel pain: a randomized controlled trial. J Orthop Sports Phys Ther. 2011 Feb;41(2):43-50. doi: 10.2519/jospt.2011.3504. Epub 2011 Jan 31. PMID 21285525
- [Background] Riddle DL, Pulisic M, Pidcoe P, Johnson RE. Risk factors for Plantar fasciitis: a matched case-control study. J Bone Joint Surg Am. 2003 May;85(5):872-7. doi: 10.2106/00004623-200305000-00015. PMID 12728038
- [Background] Martin RL, Davenport TE, Reischl SF, McPoil TG, Matheson JW, Wukich DK, McDonough CM; American Physical Therapy Association. Heel pain-plantar fasciitis: revision 2014. J Orthop Sports Phys Ther. 2014 Nov;44(11):A1-33. doi: 10.2519/jospt.2014.0303. PMID 25361863